CLINICAL TRIAL: NCT01586676
Title: Effectiveness of Motivational Interviewing Supervision in Community Programs
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Professor of Psychiatry (Psychology Section), National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: DESPR DA023230; R01DA023230 (NIH)
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2015-10

CONDITIONS: Signs and Symptoms; Clinical Supervision
Keywords: supervision; motivational interviewing; substance abuse; dissemination
MeSH Terms: conditions — Signs and Symptoms; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIA: STEP (Experimental): Motivational Interviewing Assessment: Supervisory Tools for Enhancing Proficiency (MIA: STEP)
  Interventions: Behavioral: MIA: STEP
- Supervision-as-usual (Active Comparator): Supervision-as-usual consists of the typical clinical supervision services provided to clinicians by their supervisors in their community programs.
  Interventions: Behavioral: SAU

INTERVENTIONS:
Behavioral: SAU — Supervision-as-usual
  Arms: Supervision-as-usual
Behavioral: MIA: STEP — Motivational Interviewing Assessment: Supervisory Tools for Enhancing Proficiency (MIA: STEP
  Arms: MIA: STEP

SUMMARY:
The virtual requirement that substance abuse programs use evidence-based treatments (EBT) has prompted the development of dissemination strategies to promote EBT technology transfer. Implementation research, clinical trial training methods, and clinician training studies suggest that clinical supervision that involves direct observation, fidelity rating-based feedback, and coaching of therapeutic skills is a promising dissemination approach. However, clinical supervision delivered within substance abuse programs by on-site supervisors has never been directly tested in a randomized controlled trial to determine the impact of supervision on both clinician EBT skills and client treatment outcomes.

Recent results from two NIDA CTN protocols testing the effectiveness of Motivational Interviewing (MI) have shown that community program clinicians can learn to deliver MI with fidelity when receiving MI supervision from their program supervisors after workshop training and that their implementation of MI early in treatment improves client retention and primary substance use outcomes. A MI supervision manual called MIA: STEP (Motivational Interviewing Assessment: Supervisory Tools for Enhancing Proficiency) was developed from these protocols and has begun to be widely distributed by NIDA in partnership with SAMHSA for community program use. The effectiveness of the MIA: STEP supervision approach is unknown.

This study will directly test the effectiveness of MIA: STEP supervision on clinician MI fidelity and on client outcomes by randomly assigning 60 clinicians and 420 substance-using outpatients from 11 community programs within Connecticut to one of two conditions in which clinicians in both conditions will deliver a 1-session MI intervention to clients as the enter treatment. The conditions are: 1) workshop training plus MIA: STEP supervision, and 2) workshop training alone with supervision-as-usual practices used at each program. This project will be the first randomized trial to examine the impact of clinical supervision in an empirically based treatment on both clinician and client outcomes. Moreover, because it will provide workshop training and supervision completely within the context of community programs and utilize in-house program supervisors, it will provide a rigorous evaluation of a feasible model for disseminating EBTs such as MI.

ELIGIBILITY:
For Clinicians

Inclusion Criteria:

* age 18 or older who work at one of the 12 participating programs
* willing to serve as study clinicians and learn the MI assessment intake
* working at least 20 hours per week at the program
* are not intending to give notice to their employer that they intend to leave the agency or are not scheduled for medical or family leave during the study period
* willing to record clinical sessions for review by the MI expert and/or independent raters
* willing to have supervision sessions recorded if randomized to MIA: STEP condition
* deemed capable by program administrative leadership to manage the responsibilities of being a clinician in a randomized trial

Exclusion Criteria:

* served as MI therapists in prior clinical trial studies.
* received formal supervision in MI based on direct observation, session ratings, and related feedback and coaching.
* trained as MI trainers through the Motivational Interviewing Network of Trainers (MINT).

For Clients

Inclusion Criteria:

* English-speaking
* seeking non-opiate replacement outpatient treatment for any substance use problem and have used primary substance (alcohol or illicit drug) at least once in the prior 28 days
* 18 years of age or older
* willing to participate in the protocol (randomization to clinicians contact for follow-up assessments, MI session recording for supervisor and independent review)

Exclusion Criteria:

* insufficiently medically or psychiatrically stable to participate in outpatient treatment.
* highly unlikely to be reached for follow-up due to residential instability or imminent incarceration.
* seeking detoxification only, opiate replacement treatment, or residential inpatient treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
client retention | 4-week and 12-week follow-up
  The main outcome for the client participant trial is program retention at 4-week and 12-week followups after having received a 1-session intake. Program retention is defined as the the percent days of program attendances (days attended/# days scheduled) and percent sessions attended (sessions attended/# sessions scheduled) verified by administrative record and interview with clinical staff

SECONDARY OUTCOMES:
motivational interviewing adherence and competence | baseline, post-trial and 16-weeks post-trial
  Change in clinician participant motivational interviewing (MI) adherence and competence will be measured from baseline to a post-trial point and from baseline to a 16-week post-trial follow-up point. The timeframe for the trial phase for each clinician participant will vary depending on how long it takes to be assigned and deliver the MI-base intake to 7 client participants.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Martino, Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Background] Martino S. Strategies for training counselors in evidence-based treatments. Addict Sci Clin Pract. 2010 Dec;5(2):30-9. PMID 22002451
- [Background] Olmstead TA, Abraham AJ, Martino S, Roman PM. Counselor training in several evidence-based psychosocial addiction treatments in private US substance abuse treatment centers. Drug Alcohol Depend. 2012 Jan 1;120(1-3):149-54. doi: 10.1016/j.drugalcdep.2011.07.017. Epub 2011 Aug 9. PMID 21831536
- [Background] Olmstead T, Carroll KM, Canning-Ball M, Martino S. Cost and cost-effectiveness of three strategies for training clinicians in motivational interviewing. Drug Alcohol Depend. 2011 Jul 1;116(1-3):195-202. doi: 10.1016/j.drugalcdep.2010.12.015. Epub 2011 Jan 31. PMID 21277713
- [Background] Martino S, Ball SA, Nich C, Canning-Ball M, Rounsaville BJ, Carroll KM. Teaching community program clinicians motivational interviewing using expert and train-the-trainer strategies. Addiction. 2011 Feb;106(2):428-41. doi: 10.1111/j.1360-0443.2010.03135.x. Epub 2010 Oct 6. PMID 20925684
- [Background] Martino S, Brigham GS, Higgins C, Gallon S, Freese TE, Albright LM, Hulsey EG, Krom L, Storti SA, Perl H, Nugent CD, Pintello D, Condon TP. Partnerships and pathways of dissemination: the National Institute on Drug Abuse-Substance Abuse and Mental Health Services Administration Blending Initiative in the Clinical Trials Network. J Subst Abuse Treat. 2010 Jun;38 Suppl 1(Suppl 1):S31-43. doi: 10.1016/j.jsat.2009.12.013. PMID 20307793